CLINICAL TRIAL: NCT06112093
Title: Using Repetitive Transcranial Magnetic Stimulation to Manage Headaches and Improve Rehabilitation Outcomes in Mild Traumatic Brain Injury: A Longitudinal Study
Brief Title: Repetitive Transcranial Magnetic Stimulation for Post-concussion Headaches
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Yi-Ling Kuo, PT, PhD, Assistant Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1825424
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Brain Concussion; Mild Traumatic Brain Injury; Headache; Post-Concussion Symptoms
Keywords: Repetitive transcranial magnetic stimulation; Non-invasive brain stimulation; Neuromodulation; Chronic pain; Biomarkers
MeSH Terms: conditions — Brain Concussion; Headache; Post-Concussion Syndrome; Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Moderate-dose rTMS (Active Comparator): 12 sessions (1 session/day, 3 days/week for 4 weeks) of active rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): 12 sessions (1 session/day, 3 days/week for 4 weeks) of sham rTMS will be administered at the same location and duration as the Moderate-rTMS protocol. After the study is completed, participants will be offered an opportunity to receive active rTMS.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation
- High-dose rTMS (Active Comparator): 24 sessions (4 sessions/day, 3 days/week for 2 weeks) of active rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Low-dose rTMS (Active Comparator): 6 sessions (1 session/day, 3 days/week for 2 weeks) of active rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS will be used to regulate the motor cortex to reduce headaches and post-concussion symptoms.
  Other Names: Transcranial magnetic stimulation
  Arms: High-dose rTMS; Low-dose rTMS; Moderate-dose rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation — Sham rTMS will be delivered by a sham coil as a comparator to the (active) rTMS. Sham rTMS will not change the brain function of the control group.
  Arms: Sham rTMS

SUMMARY:
This study aims to examine the long-term effect of repetitive transcranial magnetic stimulation (rTMS), a non-invasive brain stimulation technique, on chronic headaches following mild traumatic brain injury (mTBI). rTMS has been shown to be effective in reducing chronic headaches without side effects commonly seen in medications, such as sleepiness and addiction. This study uses rTMS to manage chronic headaches to improve post-concussion symptoms and reduce the economic burden due to delayed recovery. This project aims to better identify biomarkers for diagnosis and prognosis and maximize recovery from mTBI.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 55 years old
* mTBI with loss of consciousness for less than 30 min, initial Glasgow Coma Scale between 13 and 15, or post-traumatic amnesia for ≤ 24 hours
* diagnosis of persistent post-traumatic headache according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria
* headache develops within 7 days after head trauma
* headache persists for >=3 months after head trauma despite receiving standard care
* average persistent headache intensity is >= 3/10 of the numerical rating scale (NRS) on >=3days/week
* no evidence of radiculopathy or peripheral neuropathy on electromyography or clinical evaluation
* no evidence of other possible causes of headaches

Exclusion Criteria:

* history of chronic headache diagnoses such as migraine, tension, or cluster headaches prior to the incidence of mTBI
* history of other neurologic conditions with medications affecting the central nervous system
* contraindications of receiving TMS (e.g., a history of epileptic seizure and having implants like a cardiac pacemaker or intracerebral vascular clip

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2027-10-23 (Estimated)

PRIMARY OUTCOMES:
Daily headache diary | daily documentation throughout the treatment course (4 weeks)
  Composite headache score will be calculated as average intensity (NRS) × average frequency (episode/day) × average duration (hours/episode).
Patient-Reported Outcomes Measurement Information System (PROMIS) | baseline, immediately post-treatment (completion of rTMS), 1-month follow-up, 3-month follow-up, 6-month follow-up
  The PROMIS questionnaires with subsections of 1) pain interference, 2) pain behavior will be used as patient-reported outcomes of pain and sleep. For all subsections, on a scale of 1 to 5, higher numbers indicate worse outcomes.
Protein expression | baseline, immediately post-treatment (completion of rTMS)
  Peripheral blood will be collected to measure protein expression
Neurophysiological measures by TMS | baseline, immediately post-treatment (completion of rTMS)
  Neurophysiology will be measured by TMS to indicate changes in brain function.
Headache impact test 6 (HIT-6) | baseline, immediately post-treatment (completion of rTMS), 1-month follow-up, 3-month follow-up, 6-month follow-up
  The HIT-6 will be used to assess the impact of headaches on one's ability to function in occupational and social lives. On a scale of 36 to 78, higher numbers indicate worse outcomes.
Post-Concussion Symptom Scale (PCSS) | baseline, immediately post-treatment (completion of rTMS), 1-month follow-up, 3-month follow-up, 6-month follow-up
  The change in global post-concussion symptoms will be measured by the PCSS. On a scale of 1 to 5, higher numbers indicate worse outcomes.
Wrist actigraphy - physical activity level | baseline, immediately post-treatment (completion of rTMS)
  Kinematic assessments by the wrist actigraphy will be worn to measure physical activity level.
Gene expression | baseline, immediately post-treatment (completion of rTMS)
  Peripheral blood will be collected to measure mRNA to impute gene expression.

SECONDARY OUTCOMES:
Wrist actigraphy - sleep quality | baseline, immediately post-treatment (completion of rTMS)
  Kinematic assessments by the wrist actigraphy will be worn to measure sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ling Kuo, PT, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The study investigators will make the de-identified data available to users for research purposes. Sharing and modification rights of the study data will be determined for individual users by the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available no later than upon the publication of the final dataset.
Access Criteria: Study personnel on the list approved by the Institutional Review Board and researchers outside of this project as approved by the Principal Investigator

REFERENCES:
- [Background] Iverson GL, Gardner AJ, Terry DP, Ponsford JL, Sills AK, Broshek DK, Solomon GS. Predictors of clinical recovery from concussion: a systematic review. Br J Sports Med. 2017 Jun;51(12):941-948. doi: 10.1136/bjsports-2017-097729. PMID 28566342
- [Background] De Kruijk JR, Leffers P, Menheere PP, Meerhoff S, Rutten J, Twijnstra A. Prediction of post-traumatic complaints after mild traumatic brain injury: early symptoms and biochemical markers. J Neurol Neurosurg Psychiatry. 2002 Dec;73(6):727-32. doi: 10.1136/jnnp.73.6.727. PMID 12438478
- [Background] Minen MT, Boubour A, Walia H, Barr W. Post-Concussive Syndrome: a Focus on Post-Traumatic Headache and Related Cognitive, Psychiatric, and Sleep Issues. Curr Neurol Neurosci Rep. 2016 Nov;16(11):100. doi: 10.1007/s11910-016-0697-7. PMID 27709555
- [Background] Bomyea J, Lang AJ, Delano-Wood L, Jak A, Hanson KL, Sorg S, Clark AL, Schiehser DM. Neuropsychiatric Predictors of Post-Injury Headache After Mild-Moderate Traumatic Brain Injury in Veterans. Headache. 2016 Apr;56(4):699-710. doi: 10.1111/head.12799. Epub 2016 Mar 29. PMID 27028095
- [Background] Howard L, Schwedt TJ. Posttraumatic headache: recent progress. Curr Opin Neurol. 2020 Jun;33(3):316-322. doi: 10.1097/WCO.0000000000000815. PMID 32304441
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Major BP, Rogers MA, Pearce AJ. Using transcranial magnetic stimulation to quantify electrophysiological changes following concussive brain injury: a systematic review. Clin Exp Pharmacol Physiol. 2015 Apr;42(4):394-405. doi: 10.1111/1440-1681.12363. PMID 25603731
- [Background] Leung A, Shukla S, Fallah A, Song D, Lin L, Golshan S, Tsai A, Jak A, Polston G, Lee R. Repetitive Transcranial Magnetic Stimulation in Managing Mild Traumatic Brain Injury-Related Headaches. Neuromodulation. 2016 Feb;19(2):133-41. doi: 10.1111/ner.12364. Epub 2015 Nov 10. PMID 26555886
- [Background] Leung A, Fallah A, Shukla S, Lin L, Tsia A, Song D, Polston G, Lee R. rTMS in Alleviating Mild TBI Related Headaches--A Case Series. Pain Physician. 2016 Feb;19(2):E347-54. PMID 26815263
- [Background] Choi GS, Kwak SG, Lee HD, Chang MC. Effect of high-frequency repetitive transcranial magnetic stimulation on chronic central pain after mild traumatic brain injury: A pilot study. J Rehabil Med. 2018 Feb 28;50(3):246-252. doi: 10.2340/16501977-2321. PMID 29392332
- [Background] Hess JL, Tylee DS, Barve R, de Jong S, Ophoff RA, Kumarasinghe N, Tooney P, Schall U, Gardiner E, Beveridge NJ, Scott RJ, Yasawardene S, Perera A, Mendis J, Carr V, Kelly B, Cairns M; Neurobehavioural Genetics Unit; Tsuang MT, Glatt SJ. Transcriptome-wide mega-analyses reveal joint dysregulation of immunologic genes and transcription regulators in brain and blood in schizophrenia. Schizophr Res. 2016 Oct;176(2-3):114-124. doi: 10.1016/j.schres.2016.07.006. Epub 2016 Jul 20. PMID 27450777
- [Background] Hiskens MI, Schneiders AG, Angoa-Perez M, Vella RK, Fenning AS. Blood biomarkers for assessment of mild traumatic brain injury and chronic traumatic encephalopathy. Biomarkers. 2020 May;25(3):213-227. doi: 10.1080/1354750X.2020.1735521. Epub 2020 Mar 12. PMID 32096416
- [Background] Glatt SJ, Tsuang MT, Winn M, Chandler SD, Collins M, Lopez L, Weinfeld M, Carter C, Schork N, Pierce K, Courchesne E. Blood-based gene expression signatures of infants and toddlers with autism. J Am Acad Child Adolesc Psychiatry. 2012 Sep;51(9):934-44.e2. doi: 10.1016/j.jaac.2012.07.007. Epub 2012 Aug 2. PMID 22917206
- [Background] Hess JL, Quinn TP, Zhang C, Hearn GC, Chen S; Neuropsychiatric Consortium for Analysis and Sharing of Transcriptomes; Kong SW, Cairns M, Tsuang MT, Faraone SV, Glatt SJ. BrainGENIE: The Brain Gene Expression and Network Imputation Engine. Transl Psychiatry. 2023 Mar 22;13(1):98. doi: 10.1038/s41398-023-02390-w. PMID 36949060
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Askew RL, Cook KF, Revicki DA, Cella D, Amtmann D. Evidence from diverse clinical populations supported clinical validity of PROMIS pain interference and pain behavior. J Clin Epidemiol. 2016 May;73:103-11. doi: 10.1016/j.jclinepi.2015.08.035. Epub 2016 Feb 27. PMID 26931296
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Full KM, Kerr J, Grandner MA, Malhotra A, Moran K, Godoble S, Natarajan L, Soler X. Validation of a physical activity accelerometer device worn on the hip and wrist against polysomnography. Sleep Health. 2018 Apr;4(2):209-216. doi: 10.1016/j.sleh.2017.12.007. Epub 2018 Jan 17. PMID 29555136
- [Background] Kuo YL, Lin DJ, Vora I, DiCarlo JA, Edwards DJ, Kimberley TJ. Transcranial magnetic stimulation to assess motor neurophysiology after acute stroke in the United States: Feasibility, lessons learned, and values for future research. Brain Stimul. 2022 Jan-Feb;15(1):179-181. doi: 10.1016/j.brs.2021.12.001. Epub 2021 Dec 7. No abstract available. PMID 34890840
- [Background] Kuo YL, Kutch JJ, Fisher BE. Relationship between Interhemispheric Inhibition and Dexterous Hand Performance in Musicians and Non-musicians. Sci Rep. 2019 Aug 9;9(1):11574. doi: 10.1038/s41598-019-47959-y. PMID 31399612